CLINICAL TRIAL: NCT04962971
Title: Comparative Observational Study Evaluating the Urinary Comfort Related to Cystitis Symptoms Episodes and the Satisfaction of Women Following the Consumption of 3 Cranberry Extracts
Brief Title: Comparative Effect of 3 Different Cranberry Extracts on Cystitis Related Urinary Comfort in Women
Status: Completed | Type: Observational
Sponsor: CEN Biotech (Industry)
Collaborators: Nexira (Industry); CEN Nutriment (Unknown)
Responsible Party: Sponsor
Other Study IDs: C1635
Record Dates: First submitted 2021-06-17; First posted 2021-07-15 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2021-07

CONDITIONS: Recurrent Cystitis
MeSH Terms: conditions — Cystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cranberry extract X: 373 mg per Day
  Interventions: Dietary Supplement: X
- Cranberry extract Y: 404 mg per Day
  Interventions: Dietary Supplement: Y
- Cranberry extract Z: 2090 mg per Day
  Interventions: Dietary Supplement: Z

INTERVENTIONS:
Dietary Supplement: X — exocyan
  Groups: Cranberry extract X
Dietary Supplement: Y — exocyan
  Groups: Cranberry extract Y
Dietary Supplement: Z — exocyan
  Groups: Cranberry extract Z

SUMMARY:
Urinary discomfort includes a set of signs such as an urgent need to urinate, high frequency of urination per day, discomfort / difficulty or burning sensation when urinating, smelly urine. This urinary discomfort represents in women 2 to 5% of the reasons for consultation (Berg, 1991) and can have various etiologies but the bacterial origin is the most frequent. Cranberries are traditionally used for urinary comfort and the prevention of urinary disorders with bacterial origin.

The study objective is to collect in real life efficacy and tolerance data from the consumption of 3 cranberry extracts in order to highlight the qualitative and quantitative characteristics of these extracts which are directly involved in the improvement of urinary discomfort or situation of recurrent cystitis symptomatic episodes in women.

ELIGIBILITY:
Inclusion Criteria:

* having had at least 3 symptomatic episodes of cystitis (including 1 urinary tract infection confirmed by a doctor) during the last 12 months
* whose episode had a significant impact on quality of life / urinary discomfort (ACSS Dimension QoL ≥ 2)
* had a smartphone compatible with Nurstrial smartphone application (e-CRF)

Exclusion Criteria:

* to be a pregnant or breastfeeding woman or planning to be pregnant within 6 months,
* currently taking any other supplementation for urinary comfort or having taken any other cranberry-based food supplement in the past 3 months,
* to be under antibiotic treatment or during the last 7 days preceding inclusion,
* have urinary discomfort with a severe impact on quality of life (ACSS QoL> 7) during the last 24 hours prior to inclusion,
* have an allergy known to plants of the cranberry family or to one of the components of the products.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The first 216 women of the CEN Nutriment (Clinical Investigation Center) volunteer panel corresponding to the selection criteria and wishing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change of the Quality of life related to urinary discomfort | at weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  ACCS Quality of life score
Change of the Urinary comfort | on weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Visual Analogic score

SECONDARY OUTCOMES:
Intensity of urinary disconfort | Every day during each urinary symptoms episod (Week 0 to Week 24)
  Global ACCS score
Patient Global Impression of Improvement | Week 4,Week 12,Week 24
  PGI-I scale related to Urinary discomfort
Evolution of the impact of urinary discomfort on psychosocial life | Week 0,Week 4,Week 12,Week 24
  Likert 5 points scales
Duration without antibiotic treatment | on Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Collection of the intake and the duration of the antibiotic treatment, if applicable
Satisfaction of the supplementation | Week 4,Week 12,Week 24
  Likert 5 points scales
Tolerance of the supplementation | Week 4,Week 12,Week 24
  Adverse events assessment
Observance of the supplementation | on Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Total products minus remaining products

OTHER OUTCOMES:
Cystitis symptomatic episodes occurence | Week 0 to Week 24
  Number of cystitis symptomatic episodes self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Christine JUHEL, Study Director — CEN Nutriment
Locations (1):
- CEN Nutriment, Dijon, Burgundy, France

IPD SHARING:
Plan to Share IPD: Undecided